CLINICAL TRIAL: NCT06966661
Title: Peer-Supported E-Health Intervention for College Student Weight Management and Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan University Guangzhou (Other)
Collaborators: Guangzhou Sport University (Other)
Responsible Party: Principal Investigator, Ma Ruisi, Lecturer, School of Physical Education, Jinan University, Jinan University Guangzhou
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025LCLL-057
Record Dates: First submitted 2025-05-04; First posted 2025-05-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; Psychological Well Being; Obesity Prevention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (No Intervention)
- Peer Support Arm (Experimental)
  Interventions: Behavioral: Peer Support Intervention
- Peer Support eHealth Arm (Experimental)
  Interventions: Behavioral: Peer Support and eHealth Intervention

INTERVENTIONS:
Behavioral: Peer Support Intervention — In addition to all components of Standard Health Education, participants join biweekly, small-group meetings (6-8 peers) facilitated by trained upper-year student mentors who guide goal-setting, experience sharing, and mutual accountability. A moderated online chat forum provides daily encouragement, peer-to-peer Q&A, and group reminders, distinguishing this arm by its structured social support network.
  Arms: Peer Support Arm
Behavioral: Peer Support and eHealth Intervention — This arm integrates the full Peer Support Intervention with a custom mobile/web application that delivers weekly, interactive modules on nutrition, exercise, and mental health; offers in-app self-monitoring tools for weight, dietary intake, and mood; and hosts monthly live Q&A webinars with clinical nutritionists and mental health professionals. The combination of real-time peer interaction and scalable digital content differentiates it as a multifaceted, blended-delivery intervention.
  Arms: Peer Support eHealth Arm

SUMMARY:
This study will test whether adding peer support and online education can help college students manage their weight and improve their mood: we plan to enroll 300 full-time university students and randomly assign them to one of three six-month groups (monthly in-person health talks and weekly emailed tips alone; those activities plus biweekly peer-mentor meetings and an online chat group; or those activities plus a custom app delivering weekly lessons, monthly expert live Q&A, and self-tracking tools). We will measure weight, body mass index (BMI), and scores on standard questionnaires for depression (PHQ-9), anxiety (GAD-7) and life satisfaction (SWLS) at baseline, three months and six months to compare the effectiveness of each approach. By identifying which combination of face-to-face support and digital tools produces the greatest improvements, we aim to inform low-cost, scalable programs to help students maintain a healthy weight and emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* Full-time undergraduate students aged 18-25 years
* Baseline BMI ≥ 24.0 kg/m²
* Able to provide informed consent
* Owns a smartphone or computer with internet access
* Willing to attend monthly lectures and complete online modules

Exclusion Criteria:

* Current participation in another weight-management or psychological intervention program
* Diagnosis of an eating disorder, severe psychiatric illness, or medical condition affecting weight (e.g., hyperthyroidism)
* Pregnant or planning pregnancy during the study period
* Any physical limitation precluding participation in light-to-moderate physical activity
* Inability to communicate in the language of intervention materials

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 216 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | Baseline and Month 6 (6 months)
  Mean change in body weight (in kilograms) from baseline to the end of the 6-month intervention, measured by a calibrated digital scale under standardized conditions (light clothing, no shoes).

SECONDARY OUTCOMES:
Change in Depression Severity (PHQ-9) | Baseline and Month 6 (6 months)
  Mean change in Patient Health Questionnaire-9 (PHQ-9) total score from baseline to the end of the 6-month intervention. The PHQ-9 is a 9-item self-administered questionnaire used to monitor the severity of depression and response to treatment. The total score ranges from 0 to 27, where higher scores indicate greater depression severity (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- School of Physical Education, Jinan University, Guangzhou, New Territories, China

IPD SHARING:
Plan to Share IPD: Undecided
The research team will conduct in-depth analyses of key scientific questions and will maintain an embargo period to secure publication priority and preserve the integrity of the study's findings; after this period, de-identified individual participant data will be made available to qualified researchers upon request.